CLINICAL TRIAL: NCT04120168
Title: Multicenter Non-Drug Screening Study to Determine the Frequency of Duchenne Muscular Dystrophy and Late-onset Pompe Disease in Children With Unexplained Transaminase Elevation
Brief Title: Study Determining the Frequency of Duchenne Muscular Dystrophy and Late-onset Pompe Disease
Acronym: VICTORIA
Status: Completed | Type: Observational
Sponsor: Turkish Society of Pediatric Gastroenterology, Hepatology and Nutrition (Other)
Responsible Party: Sponsor
Other Study IDs: VICTORIA
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-05

CONDITIONS: Duchenne Muscular Dystrophy; Pompe Disease (Late-onset)
Keywords: CPK; Transaminase; DMD; Pompe
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Glycogen Storage Disease Type II | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — * Acid Alpha IgGlucosidase alpha enzyme test for Late Onset Pompe Disease and gene sequencing test from the same sample in samples with low enzyme activity
  * Genetic Analysis for DMD (only in boys): Detection of dystrophin gene for duplication and deletion with MLPA (Multiplex-ligation dependent probe amplification) and re-screening for other mutations by gene sequencing in patients without MLPA deletion / duplication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DMD and Pompe Disease Cohort: The aim of this study gropu was to determine the frequency of Duchenne muscular dystrophin in boys and adolescents with unexplained transaminase elevation for at least 3 months and in late onset Pompe disease in girls and boys and to determine the demographic and clinical characteristics of these patients.
  Interventions: Genetic: Laboratory Tests

INTERVENTIONS:
Genetic: Laboratory Tests — * Acid Alpha IgGlucosidase alpha enzyme test for Late Onset Pompe Disease and gene sequencing test from the same sample in samples with low enzyme activity
  * Genetic Analysis for DMD (only in boys): Detection of dystrophin gene for duplication and deletion with MLPA (Multiplex-ligation dependent probe amplification) and re-screening for other mutations by gene sequencing in patients without MLPA deletion / duplication.

SUMMARY:
This is a multicenter prospective non-drug screening study. The working period is 12 months. There is no research product to be followed or used in the study.

Demographic data, medical and family histories of the patients included in the study will be collected at the first admission. The following laboratory values of the patients will be collected:

* Alanine Transaminase (ALT)
* Aspartate Transaminase (AST)
* Gamma Glutamyl Transferase (GGT)
* Creatine Phosphokinase (CPK)
* In addition, physical examination information and Abdominal USG and Liver Biopsy Results, if any, will be collected. Following the above scans, enzyme analysis for late-onset Pompe disease in boys and girls and adolescents with high CPK levels and molecular genetic tests for Duchenne muscular dystrophy in boys and adolescents with high CPK levels will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 3 months -18 years old boys and girls
* Serum transaminase levels (serum ALT and / or AST levels> 1.52 upper limit of normal (ULN)) for at least 3 months
* The willingness of the patient and / or legal representative to sign the written consent form

Exclusion Criteria:

* Patients less than 3 months
* Patients with a known history of liver disease
* Patients with a known history of muscle disease
* Patients with a known history of rheumatologic disease
* Patients with clinical history or physical examination findings that support the possibility of liver disease (Jaundice, variceal bleeding, hepatomegaly, splenomegaly, ascites)
* ICU patients
* Patients with known congenital anomalies
* Patients with organ failure
* Patients with elevated serum GGT, Total Bliribun or Direct Bilirubin levels

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Boys and girls with unexplained transaminase elevation for at least 3 months
Sampling Method: Probability Sample
Enrollment: 590 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Frequency of Duchenne muscular dystrophin in boys and adolescents | 1 year
  The endpoints of the study were to determine the frequency of Duchenne muscular dystrophin in boys and adolescents with unexplained transaminase elevation for at least 3 months and in late onset Pompe disease in girls and boys and to determine the demographic and clinical characteristics of these patients.

CONTACTS AND LOCATIONS:
Locations (51):
- Turkey (Türkiye) (51):
  - Adana City Hospital, Adana
  - Baskent University Adana Hospital, Adana
  - Çukurova University Faculty of Medicine, Pediatric Gastroenterology, Adana
  - Afyonkarahisar Health Sciences University, Afyonkarahisar
  - Ankara Hospital, Ankara
  - Ankara University Faculty of Medicine, Pediatric Gastroenterology, Ankara
  - Ankara Yıldırım Beyazıt University, Yenimahalle Training and Research Hospital, Ankara
  - Baskent University Faculty of Medicine, Department of Pediatric Gastroenterology, Ankara
  - Gazi University Faculty of Medicine, Pediatric Gastroenterology, Ankara
  - Gülhane Training and Research Hospital, Ankara
  - Hacettepe University Faculty of Medicine, Pediatric Gastroenterology, Ankara
  - Keçiören Training and Research Hospital, Ankara
  - SBU Antalya Training and Research Hospital, Antalya
  - Bursa Yüksek İhtisas Training and Research Hospital, Bursa
  - Fatih Ünal, Bursa (Pediatric Gastroenterology Specialist), Bursa
  - Uludag University, Faculty of Medicine, Pediatric Gastroenterology, Bursa
  - Hitit University Education and Research Hospital, Çorum
  - Pamukkale University School of Medicine, Denizli
  - Fırat University Faculty of Medicine, Pediatric Gastroenterology, Elâzığ
  - Atatürk University School of Medicine, Erzurum
  - Eskisehir Osmangazi University School of Medicine, Pediatric Gastroenterology, Eskişehir
  - Gaziantep University School of Medicine, Gaziantep
  - Isparta City Hospital, Isparta
  - Süleyman Demirel University Faculty of Medicine, Isparta
  - Biruni University School of Medicine, Istanbul
  - Health Sciences University Istanbul Umraniye Health Application and Research Center, Istanbul
  - Health Sciences University Şişli Etfal Training and Research Hospital, Istanbul
  - Istanbul Altunizade Acıbadem Hospital, Istanbul
  - Istanbul Haseki Training and Research Hospital, Istanbul
  - Istanbul Medeniyet University School of Medicine, Istanbul
  - Istanbul Okmeydani Training and Research Hospital, Istanbul
  - Istinye University Faculty of Medicine, Istanbul
  - İstanbul Bakırköy Sadi Konuk Training and Research Hospital, Istanbul
  - Kanuni Sultan Süleyman Training and Research Hospital, Istanbul
  - Koç University Hospital, Istanbul
  - Marmara University School of Medicine, Pediatric Gastroenterology, Istanbul
  - Medipol University, Istanbul, Istanbul
  - Yeditepe University Faculty of Medicine, Department of Pediatric Gastroenterology, Istanbul
  - Dr. Behçet Uz Children's Hospital, Izmir
  - Health Sciences University, İzmir Tepecik Training and Research Hospital, Izmir
  - Karabuk University Faculty of Medicine, Karabük
  - Erciyes University School of Medicine, Pediatric Gasrtroenterology, Kayseri
  - Kocaeli University School of Medicine, Kocaeli
  - Selcuk University Faculty of Medicine, Pediatric Gastroenterology, Konya
  - Inonu University School of Medicine, Pediatric Gastroenterology, Malatya
  - Malatya Training and Research Hospital, Malatya
  - Mersin City Hospital, Pediatric Gastroenterology, Mersin
  - Samsun Ondokuz Mayıs University Faculty of Medicine, Samsun
  - SBU Van Regional Training and Research Hospital, Van
  - Van 100. Yıl University School of Medicine, Van
  - Bulent Ecevit University, Faculty of Medicine, Zonguldak

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kansu A, Kuloglu Z, Tumgor G, Taskin DG, Dalgic B, Caltepe G, Demiroren K, Dogan G, Tuna Kirsaclioglu C, Arslan D, Isik IA, Demir H, Bekem O, Sahin Y, Bayrak NA, Selimoglu MA, Yavuz S, Taskaya IE, Altay D; VICTORIA Study Group. The frequency of Duchenne muscular dystrophy/Becker muscular dystrophy and Pompe disease in children with isolated transaminase elevation: results from the observational VICTORIA study. Front Pediatr. 2023 Sep 25;11:1272177. doi: 10.3389/fped.2023.1272177. eCollection 2023. PMID 37818166